CLINICAL TRIAL: NCT03497130
Title: The Role of Skin Care Regimen in Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00165140
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Itching; Xerosis
Keywords: skin regimen; moisturizer; dry skin; dry; itchy skin; skin care
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regimen group (Experimental): After 1 week washout period using provided Dove® Soap without any moisturizer, participants in the skin care regimen group will receive Vaseline® Moisturizer, Dove® Soap, and application log. These participants will be asked to apply the Vaseline® Moisturizer twice a day and use Dove® Soap daily for 2 weeks. All applications should be reported in the application log by the participants. A demonstration and verbal instructions for how and where to apply the products will be provided to the subjects along with the application log for daily use.
  Interventions: Other: skin care regimen
- control group (No Intervention): After 1 week washout period using provided Dove® Soap without any moisturizer, Individuals in the control group will continue with the provided Dove® Soap for 2 weeks.
  All applications should be reported in the application log by the participants. A demonstration and verbal instructions for how and where to apply the products will be provided to the subjects along with the application log for daily use.

INTERVENTIONS:
Other: skin care regimen — These participants will be asked to apply skin care regimen, the Vaseline® Moisturizer twice a day and use Dove® Soap daily for 2 weeks.
  Arms: regimen group

SUMMARY:
This research is being done to evaluate the role of a regular skin care regimen comprising of a mild soap and moisturizer in improving dry skin and overall skin health. In this study, the investigators hope to learn the importance of regular skin care regimen in improving dry skin and overall skin health.

DETAILED DESCRIPTION:
Dry skin is a common phenomenon and can dramatically decrease a person's quality of life as well as contribute to a wide variety of skin diseases. Skin care products hydrate the skin and breaks the dry skin cycle. While there is extensive evidence of benefits of using mild cleansers and moisturizers, much of the previous studies are limited to the effects of single cleanser or moisturizer.

In this study, the investigators are going to enroll up to 100 people over the age of 18 with dry, itchy skin and they will be split into 2 groups. Participants will be randomly assigned to skin care regimen group (approximately 75% of total enrolled) and control group (approximately 25% of total enrolled). All evaluation include clinical assessments, subject questionnaires and photography will be conducted similarly in both groups.

Analysis will include paired and unpaired t-tests with two-tailed p-values. Values obtained at baseline, in middle of the study and after completing the study will be compared. The difference of measure values will be compared between application group and control group.

The moisturizing lotion and wash are generally very well tolerated.Rarely, they can induce a burning sensation, dryness, skin irritation, erythema, stinging, sensitization, and dermatitis. Risk events, problems, and deviations will be reported by the PI directly to the Institutional Review Boards.

The investigators hope to learn the importance of regular skin care regimen in improving dry skin and overall skin health.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years old with dry, itchy skin;
* Participant must be willing to comply with the requirements of the protocol;
* Participant must have the ability to understand and communicate with the investigator;
* Participant must provide informed consent.

Exclusion Criteria:

* Subjects who are unable to provide informed consent;
* Subjects who are unable to refrain from swimming or hot tub use throughout the study duration
* Subject with significant medical history or current skin diseases that the investigator feels is not safe for study participation;
* Subjects who have been treated with systemic retinoids or steroids within the past month prior to entry to the study;
* Subjects who have been treated with topical steroids, retinoids or other topical drugs within 2 weeks prior to entry to the study;
* Recently treated or current skin diseases that would affect clinical evaluation;
* Subjects who self-report that they are pregnant or nursing;
* Patients with history of investigational drug use in the 30 days prior to entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Cutaneous Translational Research Program, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawada C, Yoshida T, Yoshida H, Matsuoka R, Sakamoto W, Odanaka W, Sato T, Yamasaki T, Kanemitsu T, Masuda Y, Urushibata O. Ingested hyaluronan moisturizes dry skin. Nutr J. 2014 Jul 11;13:70. doi: 10.1186/1475-2891-13-70. PMID 25014997
- [Background] Feng L, Chandar P, Lu N, Vincent C, Bajor J, McGuiness H. Characteristic differences in barrier and hygroscopic properties between normal and cosmetic dry skin. II. Depth profile of natural moisturizing factor and cohesivity. Int J Cosmet Sci. 2014 Jun;36(3):231-8. doi: 10.1111/ics.12118. Epub 2014 Mar 29. PMID 24517532
- [Background] Rawlings AV, Harding CR. Moisturization and skin barrier function. Dermatol Ther. 2004;17 Suppl 1:43-8. doi: 10.1111/j.1396-0296.2004.04s1005.x. PMID 14728698

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen Group | Control Group
Started | 40 | 14
Completed | 39 | 13
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen Group | Control Group | Total
Number analyzed (Participants) | 40 | 14 | 54
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [24 to 53] | 24 [23 to 35] | 28 [23 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 10 | 35
  Male | 15 | 4 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 14 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Clinical Score (TCS) Between the Final Visit and Baseline
Description: Evaluated by blinded investigator, consists of three section; erythema (0=no erythema; 4=fiery red with oedema), scaling(0=no scaling; 3=severe scaling), and fissures scored 0-3 (0=no fissure; 3=wide cracks with hemorrhage) yield total between 0 and 10. The evaluation will be done for four sites: both lower legs and both forearms.Total Body Score (TCS) is the sum of three symptoms, i.e., erythema (0 = no erythema, 1 = slight erythema, 2 = moderate uniform redness, 3 = intense redness, 4 = fiery red with edema), scaling (0 = no scaling, 1 = fine scaling, 2 = moderate scaling, 3 = severe scaling with large flakes), and fissure (0 = no crack/fissure, 1 = fine cracks, 2 = single or multiple broader fissures, 3 = wide cracks with hemorrhage or exudation). Thus, the TCS could range from 0 to 10, with the higher scores representing more severe condition.
Time Frame: Baseline and 3 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Regimen Group | Control Group
Number analyzed (Participants) | 39 | 13
score on a scale | -4 [-7 to -2] | -2 [-4 to -1]

2. Primary Outcome: Change in Visual Dryness 5-point Severity Score for Total Body Score Between the Final Visit and the Baseline
Description: Visual Dryness Severity (VDS) was evaluated by blinded investigator, scored on a 5-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe, yield total between 0 and 4. The evaluation will be done for four sites: both lower legs and both forearms. Total body score is the sum of the four sites, ranging from 0 to 16 with the higher scores representing more severe dryness.
Time Frame: Baseline and 3 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Regimen Group | Control Group
Number analyzed (Participants) | 39 | 13
score on a scale | -4 [-7 to -2] | -3 [-4 to -1]

3. Secondary Outcome: Change in Frequency of Itchy-specific Quality-of-life (ItchyQoL) Score Between the Final Visit and Baseline
Description: Self-reported itchy related quality of life questions. Total 22 items and each item is scored as frequency. Frequency items are scored on scale of 1-5 (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = all the time) by four measures : Symptom with score range (6-30), Function with score range (7-35), Emotion with score range(9-45) and Overall with score range(22-110). The higher score represents more severe condition.
Time Frame: Baseline and 3 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Regimen Group | Control Group
Number analyzed (Participants) | 39 | 13
score on a scale
  symptom | -3 [-4 to -1] | 0 [-2 to 2]
  function | -1 [-3 to 0] | 0 [-2 to 2.5]
  emotion | -1 [-4 to 0] | 0 [-1.5 to 1.5]
  overall | -4 [-6 to -1] | 0 [-5.5 to 2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected within 2 weeks of product application in the study
Arm/Group | Regimen Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/13
Other Adverse Events (participants affected / at risk) | 0/39 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03497130/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03497130/ICF_001.pdf